CLINICAL TRIAL: NCT01478737
Title: A Prospective, Randomized Study on Intravitreal Ozurdex for Preventing Recurrent Vitreous Hemorrhage Following Pars Plana Vitrectomy for Proliferative Diabetic Retinopathy
Brief Title: Intravitreal Ozurdex After Pars Plana Vitrectomy for Proliferative Diabetic Retinopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Anders Kvanta (Other)
Responsible Party: Sponsor-Investigator, Anders Kvanta, Professor, St. Erik Eye Hospital
Organization: St. Erik Eye Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PDRPOZU1
Record Dates: First submitted 2011-11-21; First posted 2011-11-23 (Estimated); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Proliferative Diabetic Retinopathy
Keywords: PDRP; vitreous hemorrhage; vitrectomy
MeSH Terms: conditions — Vitreous Hemorrhage | interventions — Calcium Dobesilate; Dexamethasone; Vitrectomy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sham (Sham Comparator): Vitrectomy only
  Interventions: Procedure: Vitrectomy
- Intravitreal Ozurdex (Active Comparator): Intravitreal Ozurdex after vitrectomy
  Interventions: Drug: Intravitreal dexamethasone implant

INTERVENTIONS:
Drug: Intravitreal dexamethasone implant — Intravitreal Ozurdex after vitrectomy
  Other Names: OZURDEX® (dexamethasone intravitreal implant)
  Arms: Intravitreal Ozurdex
Procedure: Vitrectomy — Vitrectomy only
  Arms: Sham

SUMMARY:
To evaluate if intravitreal Ozurdex can reduce the incidence of recurrent vitreous hemorrhage after primary pars plana vitrectomy (PPV) in patients with proliferative diabetic retinopathy (PDRP).

DETAILED DESCRIPTION:
To perform a randomized, controlled, study on patients that undergo PPV for vitreous hemorrhage secondary to PDRP. Half of the patients will receive an intravitreal Ozurdex implant immediately after surgery. The primary outcome measure is the proportion of patients that, due to rebleeding within 12 months, have a second PPV. Secondary outcome measures include the number of episodes of vitreous hemorrhage that occur within 12 months after surgery but clear spontaneously.

ELIGIBILITY:
Inclusion Criteria:

* Patients with vitreous hemorrhage undergoing PPV for PDRP

Exclusion Criteria:

* Previous PPV
* Vitreous hemorrhage of non-PDRP origin

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-11; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Reoperation | 12 months
  The proportion of patients that, due to re-bleeding within 12 months, have a second PPV

SECONDARY OUTCOMES:
Rebleeding | 12 months
  The number of episodes of vitreous hemorrhage that occur within 12 months after surgery but clear spontaneously

CONTACTS AND LOCATIONS:
Overall Officials: Anders Kvanta, PhD, Principal Investigator — St. Erik Eye Hospital
Locations (1):
- St. Erik Eye Hospital, Stockholm, NonUS, Sweden